CLINICAL TRIAL: NCT01588808
Title: The Impact of Dietary Protein Supplementation and Age on Muscle Mass Loss During Short Term One-legged Knee Immobilization
Brief Title: Immobilization and Protein Supplementation (IM-PRO)
Acronym: IM-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Assistant Professor, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MEC 12-3-012
Record Dates: First submitted 2012-04-26; First posted 2012-05-01 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Disuse Atrophy; Aging
Keywords: Immobilization; Protein supplementation
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immobilization with protein (elderly) (Active Comparator): Immobilization with twice-daily protein supplementation - in the elderly
  Interventions: Behavioral: Immobilization
- Immobilization without protein (elderly) (Placebo Comparator): Immobilization without twice-daily protein supplementation - in the elderly
  Interventions: Behavioral: Immobilization
- Immobilization without protein (young) (Active Comparator): Immobilization without twice-daily protein supplementation - in the young
  Interventions: Behavioral: Immobilization

INTERVENTIONS:
Behavioral: Immobilization — Immobilization with protein (elderlY), immobilization without protein (elderly and young)

SUMMARY:
In the present study, the effects of 5 days of lower limb immobilization with or without twice-daily protein supplementation on muscle mass and muscle fiber characteristics will be determined. A young group will be included to compare the changes in muscle mass and muscle fiber characteristics between young and old men.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 18-35 years and from 65-75 years
* 18.5 < BMI < 30 kg/m2

Exclusion Criteria:

* Smoking
* Performing regular resistance training in the previous 6 months
* Hypertension (according to WHO criteria) [52] and/or cardiovascular disease
* Any back/leg/knee/shoulder complaints which may interfere with the use of crutches
* Systemic use of antibiotics within 3 weeks prior to the study visit
* Current systemic use of corticosteroids, growth hormone, testosterone, immunosuppressants or insulin
* Type 2 diabetes mellitus
* Any history of thrombosis
* Any family history (1st grade) of thrombosis
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Myocardial infarction within the last 3 years
* Use of anti-coagulants
* Any (history of) gastrointestinal disease that interferes with GI function
* Indications related to interaction with the study product:
* Known allergy to milk or milk products
* Known galactosemia

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | three days before immobilization, and directly after immobilization (day of cast removal; day 6)
Change in muscle fiber size | three days before immobilization, and directly after immobilization (day of cast removal; day 6)

SECONDARY OUTCOMES:
Change in muscle strength measured by quadriceps 1-Repetition Maximum by Leg Extension | Three days before immobilization, and directly after immobilization (day of cast removal; day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Dirks ML, Wall BT, Nilwik R, Weerts DH, Verdijk LB, van Loon LJ. Skeletal muscle disuse atrophy is not attenuated by dietary protein supplementation in healthy older men. J Nutr. 2014 Aug;144(8):1196-203. doi: 10.3945/jn.114.194217. Epub 2014 Jun 11. PMID 24919692